CLINICAL TRIAL: NCT06968624
Title: "Efficacy and Safety of Single Low-Dose Intravenous Ketamine for Postherpetic Neuralgia With Depression: A Randomized Controlled Study
Brief Title: Ketamine for Postherpetic Neuralgia With Depression
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-IRB202503024
Record Dates: First submitted 2025-04-25; First posted 2025-05-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Depression Disorders; Herpetic Neuralgia
Keywords: Herpetic Neuralgia; Depression; Ketamine
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine with Duloxetine (Experimental): Patients in this group received a single intravenous infusion of esketamine (esketamine at 0.2 mg/kg was added to 50 ml of normal saline and administered via a micro-infusion pump over 40 minutes), followed by 60 mg/day of oral duloxetine as maintenance therapy.
  Interventions: Drug: Intravenous Ketamine Infusions; Drug: Oral Duloxetine 60mg
- Normal saline with Duloxetine (Active Comparator): Patients in this group received a single intravenous infusion of normal saline (50 ml of normal saline administered via a micro-infusion pump over 40 minutes), followed by 60 mg/day of oral duloxetine as maintenance therapy.
  Interventions: Drug: Intravenous normal saline; Drug: Oral Duloxetine 60mg

INTERVENTIONS:
Drug: Intravenous Ketamine Infusions — The patients received a single intravenous infusion of esketamine (0.2 mg/kg), which was added to 50 ml of normal saline and administered via a micro-infusion pump over 40 minutes.
  Arms: Ketamine with Duloxetine
Drug: Intravenous normal saline — The patients received a single intravenous infusion of 50 ml normal saline via a micro-infusion pump over 40 minutes
  Arms: Normal saline with Duloxetine
Drug: Oral Duloxetine 60mg — Patients received 60 mg/day of oral duloxetine as maintenance therapy for depression.

SUMMARY:
This clinical trial examines the antidepressant efficacy and safety of a single low-dose intravenous esketamine combined with oral duloxetine in patients with postherpetic neuralgia and depression (duration more than 1 month). In this prospective, randomized, double-blind, placebo-controlled parallel study, eligible patients were randomized into two groups: one received esketamine plus duloxetine, and the other got placebo plus duloxetine. Both groups underwent standard pain management and neuro modulation therapy. The primary outcome was the Hospital Anxiety and Depression Scale - Depression( HADS-D)score at 2 weeks post - infusion, with various secondary outcomes assessed over multiple time points. Data were collected through in-person interviews and telephone follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with herpetic neuralgia, with a disease course exceeding 1 month, and an HADS-D score ≥8 (15) upon admission.
* Diagnosed with depression based on the DSM-V and ICD-11 criteria.
* Aged between 18 and 65 years old.
* BMI <30 kg/m².

Exclusion Criteria:

* Unable to cooperate with questionnaires.
* Allergic to ketamine.
* History of other mental disorders such as anxiety.
* Severe hypertension and serious dysfunctions of heart, lung, liver, or kidney.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale - Depression score | 2 weeks after intravenous ketamine infusion therapy
  This scale includes 7 items, and each item is scored from 0 to 3, so the total possible score ranges from 0 to 21. The cutoff scores usually are 0-7 for normal, 8-10 for mild, 11-14 for moderate, and 15-21 for severe depression.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale score | One day, one week, two weeks, three weeks, four weeks, five weeks and six weeks after intravenous ketamine infusion therapy
  This scale includes 10 items, each rated from 0 to 6. The total score ranges from 0 to 60. The ranges are usually 0-6 normal, 7-19 mild, 20-34 moderate, and 35-60 severe
Hospital Anxiety and Depression Scale - Anxiety score | One day, one week, two weeks, three weeks, four weeks, five weeks and six weeks after intravenous ketamine infusion therapy
  This scale includes 7 items, and each item is scored from 0 to 3, so the total possible score ranges from 0 to 21. The cutoff scores usually are 0-7 for normal, 8-10 for mild, 11-14 for moderate, and 15-21 for severe anxiety.
McGill pain score | One day, one week, two weeks, three weeks, four weeks, five weeks and six weeks after intravenous ketamine infusion therapy
  The main sections of the original MPQ are the Pain Rating Index (PRI), which includes sensory, affective, evaluative, and miscellaneous descriptors. Each category has words ranked by intensity. Then there's the Present Pain Intensity (PPI) scale, which is a 0-5 rating. Higher scores indicate more severe/intense pain
NRS( Numeric Rating Scale) pain score | One day, one week, two weeks, three weeks, four weeks, five weeks and six weeks after intravenous ketamine infusion therapy
  Rating 0-10; 0: No pain;1-3: Mild pain;4-6: Moderate pain ; 7-10: Severe pain.
Short Form-12 Quality of Life Score | One day, one week, two weeks, three weeks, four weeks, five weeks and six weeks after intravenous ketamine infusion therapy
  The Short Form-12 Health Survey (SF-12) is a widely used, self-administered questionnaire designed to assess health-related quality of life. Range: 0-100 for each component. The more scores, the better quality of life.
Columbia - Suicide Severity Rating Scale（C-SSRS）score | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a validated, clinician-administered tool designed to assess suicidal ideation and behavior.Rated on a 0-5 scale, higher scores mean higher risk of suicide.
Clinician-Administered Dissociative States Scale score | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  The Clinician-Administered Dissociative States Scale (CADSS) is a structured, clinician-administered tool designed to assess acute dissociative states in clinical and research settings. This scale includes 27 items, each item rated on a 0-4 scale, range: 0-108 .
  0-19: Minimal/no dissociation. 20-39: Mild to moderate dissociation.
  * 40: Severe dissociation (indicative of significant impairment).
Heart Rate | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  Patients' heart rate.
Peripheral capillary oxygen saturation | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  One of patients' vital signs.
Noninvasive blood pressure | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  Patients' noninvasive blood pressure
Nausea | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  Incidence of nausea after ministration of ketamine
Vomiting | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  Incidence of vomiting after administration of ketamine
Headache | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  Incidence of headache after administration of ketamine
Diplopia | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  Incidence of diplopia after administration of ketamine
Hallucination | At 2 hours and 24 hours after intravenous ketamine infusion therapy
  Incidence of hallucination after administration of ketamine

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, Phd, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: No